CLINICAL TRIAL: NCT03523559
Title: Genetic and Histopathologic Characteristics of Interstitial Cystitis
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, KYU-SUNG LEE, professor, Samsung Medical Center
Other Study IDs: 2018-03-025
Record Dates: First submitted 2018-05-01; First posted 2018-05-14 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Interstitial Cystitis
MeSH Terms: conditions — Cystitis, Interstitial

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Interstitial Cystitis
  Interventions: Genetic: bladder tissue of Interstitial Cystitis and normal bladder tissue
- normal
  Interventions: Genetic: bladder tissue of Interstitial Cystitis and normal bladder tissue

INTERVENTIONS:
Genetic: bladder tissue of Interstitial Cystitis and normal bladder tissue — Obtain the bladder tissue of Interstitial Cystitis and normal during the operation

SUMMARY:
Genetic and Histopathologic Characteristics of Interstitial Cystitis

ELIGIBILITY:
Inclusion Criteria:

* Male and female aged 19 yrs or greater
* Patients diagnosed with Hunner lesion in Interstitial cystitis and who is scheduled to undergo transurethral resection
* Patients diagnosed with Bladder cancer and who is scheduled to undergo cystectomy

Exclusion Criteria:

* Male and female under aged 20 yrs
* A person whose area of bladder cancer is larger than that of the normal area
* A person who is going to have a cystectomy after chemotherapy on bladder cancer

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Patients diagnosed with Hunner lesion in Interstitial cystitis and who is scheduled to undergo transurethral resection
  * Patients diagnosed with Bladder cancer and who is scheduled to undergo cystectomy
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2018-03-31 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Genetic differences between ulcer and non-ulcer of bladder in Interstitial Cystitis | 30days
Genetic differences between bladder tissue of Interstitial Cystitis and normal bladder tissue | 30days

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Sungkyunkwan University School of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No